CLINICAL TRIAL: NCT03674398
Title: The Efficacy of an Aerobic Exercise and Cognitive Training Program on Postconcussive Symptomology
Brief Title: Aerobic Exercise and Cognitive Training Effects on Postconcussive Symptomology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Responsible Party: Principal Investigator, Sean Mullen, Associate Professor, University of Illinois at Urbana-Champaign
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 18814
Record Dates: First submitted 2018-08-21; First posted 2018-09-17 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Post-Concussion Syndrome; Post-Traumatic Headache; Post-Concussive Syndrome, Chronic; Head Injury; MTBI - Mild Traumatic Brain Injury; Acquired Brain Injury; Closed Head Injury
Keywords: post-concussion; Mild Traumatic Brain Injury; head injury; headache; aerobic exercise; cognitive training; brain training; home-based intervention; social cognitive neuroscience
MeSH Terms: conditions — Post-Concussion Syndrome; Post-Traumatic Headache; Craniocerebral Trauma; Brain Concussion; Brain Injuries; Head Injuries, Closed; Headache

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise+CT (Experimental): Aerobic exercise for 30 minutes and smart-phone delivered cognitive training application for 20 minutes, 3 times per week for 4 weeks
  Interventions: Behavioral: Exercise+CT
- Exercise only (Active Comparator): Aerobic exercise for 30 minutes and smart-phone delivered videos for 20 minutes, 3 times per week for 4 weeks
  Interventions: Behavioral: Exercise only

INTERVENTIONS:
Behavioral: Exercise+CT — The exercise+CT group is asked to participate in 30 minutes of aerobic exercise followed by a 20-minute cognitive training (CT) program that targets attention and memory. Training will take place following exercise due to elevated levels of brain-derived neurotrophic factor and increased arousal, which is theorized to benefit cognitive task performance. Computerized CT exercises will be delivered using participants' smartphone. Adherence to the computerized CT program is monitored using electronic data upload after each training session. Participants are asked to engage in three sessions per week with the first week taking place in a lab-setting. Participants are asked to continue the aerobic exercise and CT program at home for the subsequent three weeks.
  Arms: Exercise+CT
Behavioral: Exercise only — The exercise only group will receive the same exercise prescription as the exercise+CT group. Participants in this group are asked to watch 20 minutes of health-related educational videos post-exercise. Videos are administered via participants' smartphones. After each video session, participants answer multiple-choice questions that assess engagement. Following the first week of treatment in-lab, participants are asked to continue watching health-related videos, post-exercise, for three weeks at home.
  Arms: Exercise only

SUMMARY:
The purpose of this study is to compare a 4-week, moderately intensive, lab and home-based aerobic exercise program versus exercise plus cognitive training. Participants will include individuals who experience lingering symptoms of a head injury or concussion.

DETAILED DESCRIPTION:
Eligible participants will engage in 30 minute bouts of aerobic exercise three times per week followed by a 20-minute post-exercise activity. Randomization will place participants into one of three groups: (1) aerobic exercise + cognitive training, (2) aerobic exercise + videos, or (3) waitlist control. Post-exercise activities will be delivered via participants' smartphone device by downloading the appropriate cognitive training platform or online video link.

Baseline and post-intervention assessments will consist of symptom reporting, cognitive measures, and psychosocial questionnaires. Physiological measures including heart rate and blood pressure will be assessed at baseline and at follow-up as well as during each in-lab exercise session. The wait-list control group is asked to complete all baseline and follow-up assessments and resume normal activity during the four weeks. The first week of exercise will take place in a lab-based environment, while weeks 2-4 will take place outside of the lab (participants must have access to exercise equipment at home or local fitness facility).

ELIGIBILITY:
Inclusion Criteria:

* Must have history of at least one concussion (onset was at age 18 or later)
* Ability to exercise at moderate to vigorous activity levels (defined as 50%-75% of the adjusted age-predicted maximum heart rate)
* Experiencing persistent symptoms (persistent defined as, most days per week for at least 2 weeks since sustaining injury) resulting from concussion or head injury
* Access to a smartphone and willingness to allow research staff to install application (and space to allow for installation)
* Access to a treadmill to complete exercise outside of lab environment
* Willingness to provide proof of concussion or head injury medical diagnosis
* Willingness to provide contact information of individual to confirm persistent symptoms if medical diagnosis is unavailable
* Willingness to be randomized into one of three groups

Exclusion Criteria:

* No history of concussion, head injury, or mild traumatic brain injury
* Experiencing less than 3 persistent symptoms (persistent defined as, most days per week for at least 2 weeks since sustaining injury)
* No access to a smartphone
* No access to a treadmill
* Too active (as defined by regular exercise most days per week for 30+ minutes over the past 3 months)
* Unable or unwilling to comply to lab and home-based exercise prescription
* Unable or unwilling to commit to full length of program
* Incapable of performing moderately intensive aerobic exercise OR sustaining attention to screen for 20 minutes
* Unwilling to be randomized to one of 3 groups
* Unable to commute to and from UIUC campus
* Already involved in regular weekly physical activity or cognitive training program
* Had previously diagnosed mental health condition (e.g., Major Depressive Disorder, Generalized Anxiety Disorder)
* Current involvement in litigation specific to injury

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-05-03 (Actual); Study Completion 2019-05-03 (Actual)

PRIMARY OUTCOMES:
The Rivermead Post Concussion Symptoms Questionnaire | Assessed at baseline and at 1-month follow-up
  Self reported symptoms following a head injury. Each of the 16 symptom items (e.g., sleep disturbance) is scored 0-4 (0=not experienced at all; 1=no more of a problem; 2=a mild problem; 3=a moderate problem; 4=a severe problem), yielding a total between 0 and 64. We are targeting change in total symptoms but because of the problems with "change scores" our operational definition of successful change in the primary outcome will be the time 2 total score (1-month follow-up) regressed on group while statistically adjusting for baseline score.

SECONDARY OUTCOMES:
NIH Toolbox Cognition Battery - Working Memory | Assessed at baseline and at 1-month follow-up
  List Sorting Working Memory. Participant recalls and sequences different visually and orally presented stimuli. Pictures of different foods and animals are displayed (maximum of 7 at one time) with both an accompanying audio recording and written text that name the item. Participants are asked to say the items back to the examiner in size order from smallest to largest. This test produces a standardized memory accuracy score.
NIH Toolbox Cognition Battery - Attention | Assessed at baseline and at 1-month follow-up
  Flanker Inhibitory Control and Attention. Participant focuses on a given stimulus while inhibiting attention to stimuli flanking it. Participants see a row of 5 arrows and choose the button that matches the direction the middle arrow is pointing. This test contains 20 items yielding a standardized accuracy and processing speed score.

OTHER OUTCOMES:
Psychosocial Battery - Mindfulness and Attention Awareness Scale (MAAS) | Assessed at baseline and 1-month follow-up
  Self reported items assessing experience with meditation. Participants rate 15 items on a scale from 1-6 (1=almost always; 6=almost never) yielding a mean score across the 15 items, with higher scores indicating greater mindfulness.
Psychosocial Battery - Hospital Anxiety and Depression Scale (HAD Scale) | Assessed at baseline and at 1-month follow-up
  Self reported items assessing anxiety and depression. Participants rate 14 items on a scale from 0-3 (0=not at all; 1=from time to time, occasionally; 2=a lot of the time; 3=most of the time) yielding a total score from 0-21. Three subscale scores are computed (non cases 0-7; doubtful cases 8-10; definite cases 11-21).
Cognitive Self-Efficacy - Metamemory Questionnaire (MMQ) | Assessed at baseline and at 1-month follow-up
  Self reported items assessing emotions and perceptions about current memory abilty. Participants rate 57 items on a 5-point scale (0=strongly agree/all the time; 1=agree/often; 2=undecided/sometimes; 3=disagree/rarely; 4=strongly disagree/never), yielding three subscales (contentment, ability, and strategies). Scores are added with higher scores indicating greater contentment, ability, or strategy.
Psychosocial Battery - Perceived Mental Fatigue (PMF) | Assessed at baseline, intra-session, and 1-month follow-up
  Self-reported items assessing fatigue. Participants rate their present moment feelings on a scale from 1 - 5 (1=not true at all, 5=very true) yielding a mean score across all 7 items, with higher scores indicating greater mental fatigue.

CONTACTS AND LOCATIONS:
Overall Officials: Sean P Mullen, PhD, Principal Investigator — University of Illinois at Urbana-Champaign; Daniel Palac, MA, Study Director — University of Illinois at Urbana-Champaign
Locations (1):
- University of Illinois at Urbana-Champaign, Urbana, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Although this is not an NIH-funded study, we will update these records within 1 year of data collection completion per NIH guidelines.
Access Criteria: Data will be accessible on an open site (e.g., Open Science Framework https://osf.io/) with a request to interested parties to engage with the investigative team about any publication of these data in an effort to avoid redundancy. Appropriate authorship crediting investigators involved in the parent study conceptualization, and any consultation regarding data interpretation should be sought by any researchers interested in publishing these data.

REFERENCES:
- See also: Exercise, Technology, and Cognition Laboratory — http://exercisetechlab.com